CLINICAL TRIAL: NCT02063659
Title: A Phase 3, Randomized, Placebo-controlled, Multicenter, Double-blind Study to Evaluate the Safety and Efficacy of Telotristat Etiprate (LX1606) in Patients With Carcinoid Syndrome
Brief Title: Telotristat Etiprate for Carcinoid Syndrome Therapy
Acronym: TELECAST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LX1606.1-303-CS; LX1606.303 (Other: Lexicon Pharmaceuticals, Inc.); 2013-001543-31 (EudraCT Number)
Record Dates: First submitted 2014-02-12; First posted 2014-02-14 (Estimated); Results first posted 2017-09-25 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2018-01

CONDITIONS: Carcinoid Syndrome
MeSH Terms: conditions — Serotonin Syndrome | interventions — telotristat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 250 mg Telotristat Etiprate (Experimental): Following a 3 to 4-week run-in period, participants were randomized to receive one 250 mg telotristat etiprate tablet and one placebo-matching telotristat etiprate tablet administered three times daily for 12 weeks, followed by a 36 week open-label extension period.
  Interventions: Drug: Telotristat etiprate; Drug: Placebo
- 500 mg Telotristat Etiprate (Experimental): Following a 3 to 4-week run-in period, participants were randomized to receive one 250 mg telotristat etiprate tablet and one placebo-matching telotristat etiprate tablet administered three times daily for one week, followed by two 250 mg telotristat etiprate tablets administered three times daily for 11 weeks in the 12 week double-blind treatment period, followed by a 36 week open-label extension period.
  Interventions: Drug: Telotristat etiprate; Drug: Placebo
- Placebo (Placebo Comparator): Following a 3 to 4-week run-in period, participants were randomized to receive two placebo-matching telotristat etiprate tablets administered three times daily for 12 weeks, followed by a 36 week open-label extension period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Telotristat etiprate — Telotristat etiprate tablets
  Other Names: LX1606
  Arms: 250 mg Telotristat Etiprate; 500 mg Telotristat Etiprate
Drug: Placebo — Placebo-matching telotristat etiprate tablets

SUMMARY:
The purpose of the study is to evaluate the effect of telotristat etiprate versus placebo on the incidence of treatment-emergent adverse events and on 5-hydroxyindoleacetic acid (5-HIAA) levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age
* All patients of reproductive potential must agree to use an adequate method of contraception during the study and for 12 weeks after the Follow-up visit.
* Histopathologically-confirmed, well-differentiated metastatic neuroendocrine tumor
* Documented history of carcinoid syndrome
* Patient is able and willing to provide written informed consent prior to participation

Exclusion Criteria:

* Presence of diarrhea attributed to any condition other than carcinoid syndrome.
* Presence of 12 or more watery bowel movements per day
* Positive stool examination for enteric pathogens, pathogenic ova or parasites, of Clostridium difficile at Screening
* Karnofsky Performance Status ≤ 60%
* Presence of any clinically significant laboratory, medical history, or physical examination findings deemed unacceptable by the Investigator
* A history of short bowel syndrome
* History of constipation within 2 years of Screening
* Life expectancy < 12 months from Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2014-03-11 (Actual); Primary Completion 2016-03-29 (Actual); Study Completion 2016-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Lapuerta, MD, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (45):
- United States (8):
  - Lexicon Investigational Site, Stanford, California
  - Lexicon Investigational Site, Orlando, Florida
  - Lexicon Investigational Site, Iowa City, Iowa
  - Lexicon Investigational Site, Lexington, Kentucky
  - Lexicon Investigational Site, Boston, Massachusetts
  - Lexicon Investigational Site, Buffalo, New York
  - Lexicon Investigational Site, New York, New York
  - Lexicon Investigational Site, Philadelphia, Pennsylvania
- Australia (4):
  - Lexicon Investigational Site, Kogara, New South Wales
  - Lexicon Investigational Site, St Leonards, New South Wales
  - Lexicon Investigational Site, Herston, Queensland
  - Lexicon Investigational Site, East Melbourne, Victoria
- Belgium (3):
  - Lexicon Investigational Site, Edegem
  - Lexicon Investigational Site, Ghent
  - Lexicon Investigational Site, Yvoir
- Canada (2):
  - Lexicon Investigational Site, Calgary, Alberta
  - Lexicon Investigational Site, Halifax, Nova Scotia
- France (6):
  - Lexicon Investigational Site, Clichy
  - Lexicon Investigational Site, Lille
  - Lexicon Investigational Site, Lyon
  - Lexicon Investigational Site, Marseille
  - Lexicon Investigational Site, Strasbourg
  - Lexicon Investigational Site, Villejuif
- Germany (9):
  - Lexicon Investigational Site, Bad Berka
  - Lexicon Investigational Site, Berlin
  - Lexicon Investigational Site, Hamburg
  - Lexicon Investigational Site, Heidelberg
  - Lexicon Investigational Site, Lübeck
  - Lexicon Investigational Site, Mainz
  - Lexicon Investigational Site, Marburg
  - Lexicon Investigational Site, Munich
  - Lexicon Investigational Site, Neuss
- Lexicon Investigational Site, Jerusalem, Israel
- Netherlands (3):
  - Lexicon Investigational Site, Amsterdam, North Holland
  - Lexicon Investigational Site, Noord Brahant
  - Lexicon Investigative Site, Rotterdam
- Spain (3):
  - Lexicon Investigational Site, Barcelona
  - Lexicon Investigational Site, Madrid
  - Lexicon Investigational Site, Seville
- Lexicon Investigational Site, Uppsala, Sweden
- United Kingdom (5):
  - Lexicon Investigational Site, Basingstoke Hampshire
  - Lexicon Investigational Site, Coventry
  - Lexicon Investigational Site, London
  - Lexicon Investigational Site, Manchester
  - Lexicon Investigational Site, Newcastle upon Tyne

REFERENCES:
- [Derived] Srirajaskanthan R, Pavel M, Kulke M, Clement D, Houchard A, Keeber L, Weickert MO. Weight Maintenance up to 48 Weeks in Patients With Carcinoid Syndrome Treated With Telotristat Ethyl: Pooled Data From the Open-Label Extensions of the Phase III Clinical Trials TELESTAR and TELECAST. Clin Ther. 2021 Oct;43(10):1779-1785. doi: 10.1016/j.clinthera.2021.08.014. Epub 2021 Sep 28. PMID 34598813
- [Derived] Dillon JS, Kulke MH, Horsch D, Anthony LB, Warner RRP, Bergsland E, Welin S, O'Dorisio TM, Kunz PL, McKee C, Lapuerta P, Banks P, Pavel M. Time to Sustained Improvement in Bowel Movement Frequency with Telotristat Ethyl: Analyses of Phase III Studies in Carcinoid Syndrome. J Gastrointest Cancer. 2021 Mar;52(1):212-221. doi: 10.1007/s12029-020-00375-2. PMID 32146619
- [Derived] Pavel M, Gross DJ, Benavent M, Perros P, Srirajaskanthan R, Warner RRP, Kulke MH, Anthony LB, Kunz PL, Horsch D, Weickert MO, Lapuerta P, Jiang W, Kassler-Taub K, Wason S, Fleming R, Fleming D, Garcia-Carbonero R. Telotristat ethyl in carcinoid syndrome: safety and efficacy in the TELECAST phase 3 trial. Endocr Relat Cancer. 2018 Mar;25(3):309-322. doi: 10.1530/ERC-17-0455. Epub 2018 Jan 12. PMID 29330194

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 31 investigative sites in Australia, Belgium, Canada, France, Germany, Israel, Netherlands, Spain, Sweden, United Kingdom, and the United States from 11 Mar 2014 to 29 Mar 2016.
Pre-assignment Details: Participants with Carcinoid Syndrome not adequately controlled by somatostatin analog (SSA) therapy were randomly assigned in a 1:1:1 ratio to receive placebo, 250 mg or 500 mg telotristat etiprate (LX1606) in the double-blind treatment period and were eligible to receive 500 mg telotristat etiprate in the open-label extension period.
Groups:
- Telotristat Etiprate Open-Label Extension: Patients previously assigned to 250 mg or 500 mg three times daily of telotristat etiprate were administered two 250 mg telotristat etiprate tablets three times daily in a 36 week open-label extension (OLE) period. Patients previously assigned to placebo were administered one 250 mg telotristat etiprate tablet plus one placebo-matching tablet three times daily for one week, followed by two 250 mg telotristat etiprate tablets three times daily for 35 weeks.
Period: Double-Blind Treatment Period
Arm/Group | Placebo | 250 mg Telotristat Etiprate | 500 mg Telotristat Etiprate | Telotristat Etiprate Open-Label Extension
Started | 26 | 25 | 25 | 0
Completed | 24 | 22 | 22 | 0
Not Completed | 2 | 3 | 3 | 0
Not completed — Adverse Event | 1 | 2 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Withdrawal of consent | 0 | 1 | 3 | 0
Period: Open-Label Extension Period (OLE)
Arm/Group | Placebo | 250 mg Telotristat Etiprate | 500 mg Telotristat Etiprate | Telotristat Etiprate Open-Label Extension
Started | 0 | 0 | 0 | 67
Completed | 0 | 0 | 0 | 47
Not Completed | 0 | 0 | 0 | 20
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Withdrawal of Consent | 0 | 0 | 0 | 9
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 7
Not completed — Reason not Specified | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least one dose of study drug,
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 250 mg Telotristat Etiprate | 500 mg Telotristat Etiprate | Total
Number analyzed (Participants) | 26 | 25 | 25 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (10.32) | 63.6 (12.62) | 62.7 (11.97) | 62.8 (11.52)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 12 | 14 | 15 | 41
  ≥ 65 years | 14 | 11 | 10 | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 10 | 34
  Male | 13 | 14 | 15 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 25 | 25 | 25 | 75
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 25 | 25 | 23 | 73
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 0 | 1 | 1 | 2
  Sweden | 0 | 2 | 0 | 2
  Netherlands | 3 | 2 | 1 | 6
  Belgium | 1 | 2 | 2 | 5
  United States | 4 | 5 | 7 | 16
  United Kingdom | 7 | 3 | 3 | 13
  Israel | 2 | 3 | 2 | 7
  Australia | 4 | 0 | 3 | 7
  France | 1 | 0 | 0 | 1
  Germany | 3 | 2 | 2 | 7
  Spain | 1 | 5 | 4 | 10
Somatostatin Analog (SSA) Therapy Schedule at Study Entry [Count of Participants; unit: Participants] — Patients who were on a 2-week SSA therapy or receiving SSA therapy via a subcutaneous continuous infusion pump are included in the "4-week" category.
  Participants
    3-Week | 6 | 7 | 9 | 22
    4-Week | 20 | 15 | 11 | 46
    Not on SSA | 0 | 3 | 5 | 8
SSA Therapy Name at Study Entry [Count of Participants; unit: Participants]
  Octreotide | 12 | 17 | 16 | 45
  Lanreotide | 14 | 5 | 3 | 22
  Unknown | 0 | 0 | 1 | 1
  Not Applicable | 0 | 3 | 5 | 8
Childbearing Potential [Count of Participants; unit: Participants]
  Yes | 2 | 4 | 1 | 7
  No | 11 | 7 | 9 | 27
  Not Applicable | 13 | 14 | 15 | 42
Urinary 5-Hydroxyindoleacetic acid (5-HIAA) at Randomization [Count of Participants; unit: Participants] — ULN=upper limit of normal.
  Participants
    ≤ ULN | 9 | 5 | 8 | 22
    > ULN | 17 | 18 | 17 | 52
    Unknown | 0 | 2 | 0 | 2
Region [Count of Participants; unit: Participants]
  North America | 4 | 6 | 8 | 18
  Europe | 16 | 16 | 12 | 44
  Rest of the World | 6 | 3 | 5 | 14
Weight [Mean (Standard Deviation); unit: kg] | 76.38 (16.959) | 74.74 (17.839) | 76.69 (26.188) | 75.94 (20.442)
Height [Mean (Standard Deviation); unit: cm] | 169.48 (9.765) | 169.74 (10.025) | 170.08 (8.525) | 169.76 (9.327)
Baseline Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI was calculated by weight (kg) / (height [cm] × 0.01)^2.
  kg/m^2 | 26.28 (4.364) | 25.96 (5.258) | 26.21 (9.213) | 26.16 (6.521)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) in the Double-Blind Treatment Period
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. A TEAE was an AE reported after the first dose of randomized treatment on Day 1.
Time Frame: First dose of study drug to within 30 days of last dose of study drug in the Double-Blind Treatment Period (Up to 17.1 Weeks)
Population: Safety population, defined as all participants who received at least one dose of study drug, was used for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 250 mg Telotristat Etiprate | 500 mg Telotristat Etiprate
Number analyzed (Participants) | 26 | 25 | 25
Participants | 21 | 25 | 22

2. Primary Outcome: Primary: Percent Change From Baseline in Urinary 5-hydroxyindoleacetic Acid (u5-HIAA) Levels
Description: u5-HIAA is a standard test used in clinical practice to assess neuroendocrine tumor (NET) activity and is collected as a 24-hour urine specimen. A negative change from Baseline indicates improvement.
Time Frame: Baseline and 12 Weeks
Population: Participants from the Intent-to-treat population, all randomized participants, with data available for this endpoint were included in the analysis.
Measure: Mean (Standard Deviation); unit: percentage change of mg/24 hours
Arm/Group | Placebo | 250 mg Telotristat Etiprate | 500 mg Telotristat Etiprate
Number analyzed (Participants) | 22 | 17 | 19
percentage change of mg/24 hours | 97.721 (397.0107) | -33.164 (58.4754) | -76.466 (17.3714)
Statistical Analysis 1: Comparison: Placebo vs 250 mg Telotristat Etiprate; The primary analysis used a blocked 2-sample Wilcoxon rank sum statistic stratified by the u5-HIAA at randomization; Test type: Superiority; p < 0.001, Wilcoxon rank sum; Hodges-Lehman estimator of difference = -53.955, 95% CI 2-sided [-84.955 to -25.119]; Mean difference is calculated as LX1606-Placebo
Statistical Analysis 2: Comparison: Placebo vs 500 mg Telotristat Etiprate; The primary analysis used a blocked 2-sample Wilcoxon rank sum statistic stratified by the u5-HIAA at randomization; Test type: Superiority; p < 0.001, Wilcoxon rank sum; Hodges-Lehman estimator of difference = -89.662, 95% CI 2-sided [-113.104 to -63.863]; Mean difference is calculated as LX1606-Placebo

3. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) in the Open-Label Extension Period
Description: as for outcome 1
Time Frame: First dose of study drug to within 30 days of last dose of study drug in the Open-Label Extension Period (Up to 52.6 Weeks)
Population: Safety population, defined as all participants who received at least one dose of study drug, was used for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Telotristat Etiprate Open-Label Extension
Number analyzed (Participants) | 67
Participants | 61

4. Secondary Outcome: Change From Baseline in the Number of Bowel Movements (BMs) Per Day Averaged Over 12 Weeks
Description: Participants recorded the number of bowel movements per day in a daily diary. The total number of BMs per day were averaged over the 12-week period. A negative change from Baseline indicates improvement.
Time Frame: Baseline and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: counts/day
Arm/Group | Placebo | 250 mg Telotristat Etiprate | 500 mg Telotristat Etiprate
Number analyzed (Participants) | 25 | 25 | 25
counts/day | 0.050 (0.3263) | -0.452 (0.6940) | -0.595 (0.7240)

5. Secondary Outcome: Change From Baseline in Stool Form/Consistency Averaged Across All Time-Points
Description: Participants assessed stool form/consistency of a BM using the Bristol Stool Form Scale where: 1=hard lumps to 7=watery liquid. The daily scores were averaged over the 12-week period. A negative change indicates improvement.
Time Frame: Baseline and 12 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | 250 mg Telotristat Etiprate | 500 mg Telotristat Etiprate
Number analyzed (Participants) | 25 | 25 | 25
score on a scale | 0.006 (0.4127) | -0.196 (0.7012) | -0.597 (0.8605)

6. Secondary Outcome: Change From Baseline in the Number of Daily Cutaneous Flushing Episodes Averaged Across All Time-Points
Description: Participants recorded the number daily flushing episodes per day in a daily diary. The total number of flushing episodes per day were averaged over the 12-week period. A negative change from Baseline indicates improvement.
Time Frame: Baseline and 12 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: counts/day
Arm/Group | Placebo | 250 mg Telotristat Etiprate | 500 mg Telotristat Etiprate
Number analyzed (Participants) | 25 | 25 | 25
counts/day | -0.333 (1.2203) | -0.061 (0.9754) | 0.114 (2.0992)

7. Secondary Outcome: Change From Baseline in Abdominal Pain Averaged Across All Time-Points
Description: Participants recorded abdominal pain in a daily diary. Participants evaluated the level of any abdominal pain using an 11-point numeric rating scale, where: 0=no pain to 10=worst pain ever experienced. The average daily abdominal pain was averaged over the 12-week period. A negative change from Baseline indicates improvement.
Time Frame: Baseline and 12 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | 250 mg Telotristat Etiprate | 500 mg Telotristat Etiprate
Number analyzed (Participants) | 25 | 25 | 25
score on a scale | -0.063 (0.7823) | -0.234 (0.9697) | 0.025 (0.7744)

8. Secondary Outcome: Change in the Frequency of Rescue Short-acting, Somatostatin Analog (SSA) Used to Treat Carcinoid Syndrome Symptoms Averaged Across All Time-Points
Description: The frequency (the number of times) the participant used rescue with SSA to control symptoms was recorded in a daily diary. The daily number of rescue treatments with SSA was averaged over the 12- week period. A negative change from Baseline (less use of SSA) indicates improvement.
Time Frame: Baseline and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: counts/day
Arm/Group | Placebo | 250 mg Telotristat Etiprate | 500 mg Telotristat Etiprate
Number analyzed (Participants) | 25 | 25 | 25
counts/day | -0.013 (0.1359) | -0.065 (0.3542) | 0.006 (0.1030)

9. Secondary Outcome: Change From Baseline in the Number of Daily BMs Averaged Over the 12-Week Double-Blind Period, Among Participants Who Were Not Receiving SSA Therapy at Baseline
Description: as for outcome 4
Time Frame: Baseline and 12 Weeks
Population: Participants from the Intent-to-treat population, all randomized participants, with data available for this endpoint were included in the analysis.The Placebo arm is not included because all participants in the Placebo arm were receiving SSA therapy at Baseline.
Measure: Mean (Standard Deviation); unit: counts/day
Arm/Group | 250 mg Telotristat Etiprate | 500 mg Telotristat Etiprate
Number analyzed (Participants) | 3 | 5
counts/day | -0.906 (0.5925) | -0.98 (1.154)

ADVERSE EVENTS:
Time Frame: First dose of study drug to within 30 days of last dose of study drug (Up to 77.7 Weeks)
Description: Data for the double-blind treatment period and the open-label extension period were analyzed separately. In the Non-Serious Adverse Event section, a result of "0" for a preferred term means that there are no participants in that arm above the 5% threshold.
Arm/Group | Placebo | 250 mg Telotristat Etiprate | 500 mg Telotristat Etiprate | Telotristat Etiprate Open-Label Extension
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/25 | 0/25 | 0/67
Serious Adverse Events (participants affected / at risk) | 5/26 | 1/25 | 3/25 | 17/67
Other Adverse Events (participants affected / at risk) | 21/26 | 25/25 | 22/25 | 61/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=26) | 250 mg Telotristat Etiprate (N=25) | 500 mg Telotristat Etiprate (N=25) | Telotristat Etiprate Open-Label Extension (N=67)
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Urethral stent insertion (Surgical and medical procedures) | 1 | 0 | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 0 | 0 | 0
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wound secretion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Diagnostic procedure (Investigations) | 0 | 0 | 0 | 1
Hepatectomy (Surgical and medical procedures) | 0 | 0 | 0 | 2
Small intestinal resection (Surgical and medical procedures) | 0 | 0 | 0 | 2
Antibiotic prophylaxis (Surgical and medical procedures) | 0 | 0 | 0 | 1
Therapeutic embolisation (Surgical and medical procedures) | 0 | 0 | 0 | 1
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 3
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Herpes zoster ophthalmic (Infections and infestations) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=26) | 250 mg Telotristat Etiprate (N=25) | 500 mg Telotristat Etiprate (N=25) | Telotristat Etiprate Open-Label Extension (N=67)
Abdominal pain (Gastrointestinal disorders) | 4 | 8 | 1 | 12
Diarrhoea (Gastrointestinal disorders) | 5 | 4 | 2 | 9
Nausea (Gastrointestinal disorders) | 4 | 3 | 2 | 14
Constipation (Gastrointestinal disorders) | 1 | 4 | 3 | 8
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1 | 2 | 5
Abdominal distension (Gastrointestinal disorders) | 0 | 3 | 1 | 4
Dyspepsia (Gastrointestinal disorders) | 2 | 2 | 0 | 0
Fatigue (General disorders) | 2 | 3 | 2 | 7
Asthenia (General disorders) | 2 | 1 | 0 | 7
Oedema peripheral (General disorders) | 0 | 2 | 1 | 5
Pyrexia (General disorders) | 0 | 3 | 0 | 6
Urinary tract infection (Infections and infestations) | 0 | 3 | 0 | 0
Influenzae (Infections and infestations) | 0 | 0 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Dizziness (Nervous system disorders) | 3 | 0 | 2 | 0
Depressed mood (Psychiatric disorders) | 2 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0
Flushing (Vascular disorders) | 2 | 3 | 0 | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 4
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 4
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 4
Weight decreased (Investigations) | 0 | 0 | 0 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 4
Headache (Nervous system disorders) | 0 | 0 | 0 | 5
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 5
Depression (Psychiatric disorders) | 0 | 0 | 0 | 8
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution must provide any proposed publication or presentation to Sponsor for Sponsor's review, comment and approval at least thirty (30) days prior to the proposed submission for publication date or the proposed presentation date. Sponsor shall have the right to have deleted from the final version of the publication any Confidential Information, proprietary information or patentable subject matter.